CLINICAL TRIAL: NCT06496243
Title: A Phase 2 Study to Evaluate the Effect of Obicetrapib Alone and in Combination With Evolocumab (Repatha®) on Lipoprotein (a) in Patients With Mild Dyslipidemia: The VINCENT Study
Brief Title: Impact of Obicetrapib and Obicetrapib Plus Repatha on Lp(a) Levels
Acronym: VINCENT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TA-8995-206
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-05

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: 8 weeks on 10 mg daily obicetrapid followed by 8 weeks on obicetrapib 10 mg daily/Repatha 140 mg SC every 2 weeks combination therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- obicetrapib/evolocumab combination (Experimental): obicetrapib 10 mg/dL daily for 8 weeks followed by obicetrapib 10 mg/dL daily + evolocumab 140 mg/dL every other week for 8 weeks
  Interventions: Drug: obicetrapib 10 mg + obicetrapib/evolocumab 140 mg Q 2 weeks

INTERVENTIONS:
Drug: obicetrapib 10 mg + obicetrapib/evolocumab 140 mg Q 2 weeks — 10 mg obicetrapib for 8 weeks followed by 10 mg obicetrapib/ 140 mg evolocumab (every 2 weeks) combination for 8 weeks
  Other Names: Repatha

SUMMARY:
The goal of this open label 16 week trial is to evaluate Lp(a) levels for patients with elevated Lp(a) being treated with obicetrapib and obiceptrapib/evolocumab

Patients will:

Have baseline Lp(a) tested at randomization Take 10mg/dL obiceptrapib daily for 8 weeks and have Lp(a) tested at Week 8 Take 10 mg/dL obicetrapib daily/evolocumab 140 every other week for 8 weeks and have Lp(a) retested at Week 16

ELIGIBILITY:
Inclusion Criteria:

* Lp(a): >=50 mg/dL (>=125 nmol/L) for cohort 1 (FILLED) and Lp(a) >= 20 mg/dL (>= 50 nmol/L) to <50 mg/dL (< 125 nmol/L) for cohort 2
* LDL-C >70 mg/dL
* TG < 400mg/dL (<4.52 mmol/L)

Exclusion Criteria:

* HbA1c>=10 or FPG >=270 mg/dL
* CV events within 3 months of screen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of evolocumab in combination with obicetrapib on lipoprotein (a) (Lp[a]). | 16 weeks from baseline; 8 weeks on combination therapy
  Lp(a) change on combination therapy

SECONDARY OUTCOMES:
To evaluate the effect of obicetrapib alone on Lp(a). | 8 weeks
  Lp(a) change on obicetrapib

CONTACTS AND LOCATIONS:
Locations (1):
- UPenn, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No